CLINICAL TRIAL: NCT02616484
Title: Phase 3 Trial of Dichloroacetate in Pyruvate Dehydrogenase Complex Deficiency:
Brief Title: Trial of Dichloroacetate in Pyruvate Dehydrogenase Complex Deficiency:
Acronym: DCA/PDCD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Saol Therapeutics Inc (Industry)
Collaborators: Medosome Biotec LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB201500698 - A - N
Record Dates: First submitted 2015-11-17; First posted 2015-11-30 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Pyruvate Dehydrogenase Complex Deficiency
Keywords: Sodium Dichloroacetate; Treatment of PDCD with Dichloroacetate
MeSH Terms: conditions — Pyruvate Dehydrogenase Complex Deficiency Disease | interventions — Dichloroacetic Acid; Genotype

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dichloroacetate, then Placebo (Active Comparator): This group will start on the Dichloroacetate (DCA) treatment which will last for 4 months. After 4 months a 1 month washout period will occur. After the 1 month the group will crossover to the placebo treatment for 4 months.
  Participants will be genotyped to determine GSTZ1 (glutathione S-transferase Zeta-1) haplotype status, which will stratify this group into 1 of 2 dose regimens
  Interventions: Drug: Dichloroacetate (DCA); Other: Placebo; Genetic: Genotype
- Placebo, then Dichloroacetate (Placebo Comparator): This group will start on the placebo treatment which will last for 4 months. After 4 months a 1 month washout period will occur. After the 1 month the group will crossover to the Dichloroacetate (DCA) treatment for 4 months.
  Participants will be genotyped to determine GSTZ1 (glutathione S-transferase Zeta-1) haplotype status, which will stratify this group into 1 of 2 dose regimens
  Interventions: Drug: Dichloroacetate (DCA); Other: Placebo; Genetic: Genotype

INTERVENTIONS:
Drug: Dichloroacetate (DCA) — Study medication DCA is an oral solution mixed with an artificial sweetener containing aspartame and strawberry extract (50mg/mL)
  Participants will be genotyped to determine GSTZ1 (glutathione S-transferase Zeta-1) haplotype status, which will stratify this group into 1 of 2 dose regimens:
  EGT carriers will receive 12 mg/kg/12hr DCA. EGT non-carriers will receive 6 mg/kg/12 hr DCA.
  Other Names: Sodium Dichloroacetate
Other: Placebo — Participants will receive the same volume of placebo in liquid form given during DCA treatment arm. Liquid will be an exact replication of DCA formulation with no DCA added.
Genetic: Genotype — Participants will be genotyped to determine GSTZ1 haplotype status.

SUMMARY:
The objective of this research study is to conduct a pivotal phase 3 trial of treatment with the investigational drug dichloroacetate (DCA) in young children with deficiency of the pyruvate dehydrogenase complex (PDC). PDC deficiency (PDCD) is the most common cause of congenital lactic acidosis and is a frequently fatal metabolic disease of childhood for which no proven treatment exists. The investigators predict that DCA represents targeted potential therapy for PDCD because of its ability to increase both the catalytic activity and stability of the enzyme complex. The conclusions of numerous laboratory and clinical investigations are consistent with this postulate and have led to the designation of DCA as an Orphan Product for congenital lactic acidosis by the Food and Drug Administration.

A novel Observer reported outcome (ObsRO) survey that is completed by study participant's parent/caregiver, is the efficacy outcome measure.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
Clinical sites will be established across the United States for study participation. The investigators will conduct a randomized, placebo-controlled, double-blind trial of 24 evaluable children (30 randomized), aged 6 months through 17 years, with confirmed diagnosis of PDC Deficiency.

Study participants complete Screening procedures at Visit 1 to confirm eligibility for study participation. Screening study procedures include medical history review and physical exam; blood and urine collection, and collection of cheek (buccal) cells; training to complete the ObsRO daily survey. The ObsRO is a survey developed for this study to evaluate how study participants are feeling and functioning in the home setting. The ObsRO survey is completed by the study participant parent/caregiver every day during both treatment periods (study medication and placebo) of study participation (approximately 9 months). During treatment period 1 and 2 (4 months of study medication and 5 months of placebo), the study participant will communicate with the study team at least 2 times per month to evaluate the child's level of health, and compliance with daily survey completion and taking the study medication.

Study participants complete Baseline study procedures at Visit 2 prior to randomization to treatment. Baseline study procedures include, medical history review and physical exam; blood and urine collection; 3 day food record. The study medication will be shipped to the study participants home each month of study participation.

Safety labs are completed during each randomization period (month 3 and month 5). The safety labs can be completed at the clinical trial site, or at any standard clinical laboratory.

Study participants will complete a study visit after each randomization period (month 5 and 9) to complete study assessments at the same clinical site. Visit study procedures include medical history review and physical exam; blood and urine collection; 3 day food record.

Study participants who complete both treatment periods and did not sustain serious adverse events attributable to DCA, will be offered continued access to investigational medication DCA through an open-label access program until the study concludes. Study participants must sign a separate consent form for participation in the open-label access phase of this clinical trial and must complete a study visit every 6 months at the same clinical site for study assessments that include medical history review and physical exam, blood and urine collection. The study medication will continue to be mailed to the study participant during the open-label phase at the same dose received during the blinded phase of the study.

Study participants will be stratified according to their predicted rate of DCA metabolism and clearance, based on genotyping prior to randomization (completed at visit 1 buccal cell collection).

Study participants will continue whatever diet and other "standard of care" is deemed appropriate by their local expert clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 m through 17 y
* Presence of characteristic clinical or metabolic features of pyruvate dehydrogenase complex deficiency (PDCD) and
* Presence of a known pathogenic mutation of a gene that is specifically associated with PDCD.

Exclusion Criteria:

A genetic mitochondrial disease other than those stipulated under inclusion criteria Primary disorders of amino acid metabolism; primary disorders of fatty acid oxidation Secondary lactic acidosis due to impaired oxygenation or circulation (cardiomyopathy or congenital heart defect) Renal insufficiency (defined as: requires chronic dialysis or serum creatinine ≥ 1.2 mg/dl; creatinine clearance <60 ml/min Primary hepatic disease unrelated to PDCD Pregnancy or breast feeding

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2025-08-27 (Estimated); Study Completion 2025-08-27 (Estimated)

PRIMARY OUTCOMES:
The efficacy will be measured between the groups by using the Observer Reported Outcome (ObsRO) measure of health. | 9 months
  The efficacy of dichloroacetate will be determined by applying a novel Observer Reported Outcome (ObsRO) measure of health. The ObsRO scores will be graded on a Likert Scale from 0-4. (0 being absent and 4 being extremely severe).
The number of participants with adverse events will be compared between the groups. | 9 months
  This is to evaluate the safety and tolerability of dichloroacetate by comparing the 1) number and 2) severity of adverse events during both the double-blind and open label treatment phases.

SECONDARY OUTCOMES:
Karnofsky/Lansky Performance Status | 9 months
  The Karnofsky/Lansky performance Scale is completed by the study team. It is a measure of the study participants functional ability to carry on activities of daily living.
  The Karnofsky Scale is used for study participants age greater than 16 years. The Lansky Scale is used for study participants age less than 16 years.
Blood lactate levels between the groups. | 9 months
  The measurement of blood lactate level will be performed.
Plasma β-hydroxybutyrate (β-OHB) concentrations between the groups. | 9 months
  The measurement of plasma β-hydroxybutyrate (β-OHB) concentrations will be performed.

OTHER OUTCOMES:
The number of participants with adverse events based on the age at randomization between the groups. | 9 months
  The number of participants with adverse events based on the age at randomization will be measured between the groups.
The number of participants with adverse events based on dietary fat intake between the groups. | 9 months
  The number of participants with adverse events based on dietary fat intake will be measured between the groups.
The efficacy will be measured using the Observer Reported Outcome (ObsRO) scale of health based on the genetic-based dosing between the groups. | 9 months
  The efficacy of dichloroacetate will be determined by using the Observer Reported Outcome (ObsRO) measure of health based on the GSTZ1 haplotype status, genetic-based dosing. The ObsRO scores will be graded on a Likert Scale from 0-4. (0 being absent and 4 being extremely severe).
The efficacy will be measured using the Observer Reported Outcome (ObsRO) scale of health based on the age at randomization between the groups | 9 months
  The efficacy of dichloroacetate will be determined by using the Observer Reported Outcome (ObsRO) measure of health based on the age at randomization. The ObsRO scores will be graded on a Likert Scale from 0-4. (0 being absent and 4 being extremely severe).
The efficacy will be measured using the Observer Reported Outcome (ObsRO) scale of health based on the dietary fat intake between the groups | 9 months
  The efficacy of dichloroacetate will be determined by using the Observer Reported Outcome (ObsRO) measure of health based on the dietary fat intake. The ObsRO scores will be graded on a Likert Scale from 0-4. (0 being absent and 4 being extremely severe).

CONTACTS AND LOCATIONS:
Overall Officials: Richard Neibeger, MD, Principal Investigator — University of Florida
Locations (10):
- United States (10):
  - Children's Hospital of Orange County, Orange, California
  - Stanford University, Stanford, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel KP, O'Brien TW, Subramony SH, Shuster J, Stacpoole PW. The spectrum of pyruvate dehydrogenase complex deficiency: clinical, biochemical and genetic features in 371 patients. Mol Genet Metab. 2012 Jul;106(3):385-94. doi: 10.1016/j.ymgme.2012.03.017. PMID 22896851
- [Background] DeBrosse SD, Okajima K, Zhang S, Nakouzi G, Schmotzer CL, Lusk-Kopp M, Frohnapfel MB, Grahame G, Kerr DS. Spectrum of neurological and survival outcomes in pyruvate dehydrogenase complex (PDC) deficiency: lack of correlation with genotype. Mol Genet Metab. 2012 Nov;107(3):394-402. doi: 10.1016/j.ymgme.2012.09.001. Epub 2012 Sep 7. PMID 23021068
- [Background] Ferriero R, Manco G, Lamantea E, Nusco E, Ferrante MI, Sordino P, Stacpoole PW, Lee B, Zeviani M, Brunetti-Pierri N. Phenylbutyrate therapy for pyruvate dehydrogenase complex deficiency and lactic acidosis. Sci Transl Med. 2013 Mar 6;5(175):175ra31. doi: 10.1126/scitranslmed.3004986. PMID 23467562
- [Background] Stacpoole PW. The dichloroacetate dilemma: environmental hazard versus therapeutic goldmine--both or neither? Environ Health Perspect. 2011 Feb;119(2):155-8. doi: 10.1289/ehp.1002554. Epub 2010 Oct 4. PMID 20920954
- [Background] Evans OB, Stacpoole PW. Prolonged hypolactatemia and increased total pyruvate dehydrogenase activity by dichloroacetate. Biochem Pharmacol. 1982 Apr 1;31(7):1295-300. doi: 10.1016/0006-2952(82)90019-3. PMID 7092922
- [Background] Han Z, Berendzen K, Zhong L, Surolia I, Chouthai N, Zhao W, Maina N, Srivastava A, Stacpoole PW. A combined therapeutic approach for pyruvate dehydrogenase deficiency using self-complementary adeno-associated virus serotype-specific vectors and dichloroacetate. Mol Genet Metab. 2008 Apr;93(4):381-7. doi: 10.1016/j.ymgme.2007.10.131. Epub 2008 Feb 21. PMID 18206410
- [Background] Ishida N, Kitagawa M, Hatakeyama S, Nakayama K. Phosphorylation at serine 10, a major phosphorylation site of p27(Kip1), increases its protein stability. J Biol Chem. 2000 Aug 18;275(33):25146-54. doi: 10.1074/jbc.M001144200. PMID 10831586
- [Background] Lu KP, Liou YC, Zhou XZ. Pinning down proline-directed phosphorylation signaling. Trends Cell Biol. 2002 Apr;12(4):164-72. doi: 10.1016/s0962-8924(02)02253-5. PMID 11978535
- [Background] Virshup DM, Eide EJ, Forger DB, Gallego M, Harnish EV. Reversible protein phosphorylation regulates circadian rhythms. Cold Spring Harb Symp Quant Biol. 2007;72:413-20. doi: 10.1101/sqb.2007.72.048. PMID 18419299
- [Background] Moretto-Zita M, Jin H, Shen Z, Zhao T, Briggs SP, Xu Y. Phosphorylation stabilizes Nanog by promoting its interaction with Pin1. Proc Natl Acad Sci U S A. 2010 Jul 27;107(30):13312-7. doi: 10.1073/pnas.1005847107. Epub 2010 Jul 9. PMID 20622153
- [Background] Thomas LW, Lam C, Edwards SW. Mcl-1; the molecular regulation of protein function. FEBS Lett. 2010 Jul 16;584(14):2981-9. doi: 10.1016/j.febslet.2010.05.061. Epub 2010 Jun 11. PMID 20540941
- [Background] Henderson GH, Whalen PO, Darr RA, Curry SH, Derendorf H, Baumgartner TG, Stacpoole PW: Development of an oral drug formulation for dichloroacetate and thiamine. Drug Devel Indust Pharm, 20:2425-2437, 1994.
- [Background] Chu PI, Curry SH, Baumgartner TG, Henderson GN, Stacpoole PW. Preparation and stability of intravenous solutions of sodium dichloroacetate (DCA). J Parenter Sci Technol. 1992 Jan-Feb;46(1):16-8. PMID 1625103
- [Background] Berendzen K, Theriaque DW, Shuster J, Stacpoole PW. Therapeutic potential of dichloroacetate for pyruvate dehydrogenase complex deficiency. Mitochondrion. 2006 Jun;6(3):126-35. doi: 10.1016/j.mito.2006.04.001. Epub 2006 May 3. PMID 16725381
- [Background] Stacpoole PW, Kerr DS, Barnes C, Bunch ST, Carney PR, Fennell EM, Felitsyn NM, Gilmore RL, Greer M, Henderson GN, Hutson AD, Neiberger RE, O'Brien RG, Perkins LA, Quisling RG, Shroads AL, Shuster JJ, Silverstein JH, Theriaque DW, Valenstein E. Controlled clinical trial of dichloroacetate for treatment of congenital lactic acidosis in children. Pediatrics. 2006 May;117(5):1519-31. doi: 10.1542/peds.2005-1226. PMID 16651305
- [Background] Stacpoole PW, Gilbert LR, Neiberger RE, Carney PR, Valenstein E, Theriaque DW, Shuster JJ. Evaluation of long-term treatment of children with congenital lactic acidosis with dichloroacetate. Pediatrics. 2008 May;121(5):e1223-8. doi: 10.1542/peds.2007-2062. Epub 2008 Apr 14. PMID 18411236
- [Background] Abdelmalak M, Lew A, Ramezani R, Shroads AL, Coats BS, Langaee T, Shankar MN, Neiberger RE, Subramony SH, Stacpoole PW. Long-term safety of dichloroacetate in congenital lactic acidosis. Mol Genet Metab. 2013 Jun;109(2):139-43. doi: 10.1016/j.ymgme.2013.03.019. Epub 2013 Apr 6. PMID 23611579
- [Background] Robinson BH. Lactic academia (disorders of pyruvate carboxylase, pyruvate dehydrogenase). In: Scriver CR, Beaudet AL, Sly WS, Valle D. (Eds.). The metabolic and molecular bases of inherited disease, seventh ed. McGraw-Hill, New York, pp. 1479-1499, 1995.
- [Background] Ozlu N, Akten B, Timm W, Haseley N, Steen H, Steen JAJ. Phosphoproteomics. Wiley Interdiscip Rev Syst Biol Med. 2010 May-Jun;2(3):255-276. doi: 10.1002/wsbm.41. PMID 20836028
- [Background] U.S. Department of Health and Human Services FDA Center for Drug Evaluation and Research; U.S. Department of Health and Human Services FDA Center for Biologics Evaluation and Research; U.S. Department of Health and Human Services FDA Center for Devices and Radiological Health. Guidance for industry: patient-reported outcome measures: use in medical product development to support labeling claims: draft guidance. Health Qual Life Outcomes. 2006 Oct 11;4:79. doi: 10.1186/1477-7525-4-79. PMID 17034633
- [Background] Papadopoulos EJ, Patrick DL, Tassinari MS, Mulberg AE, Epps C, Pariser AR, Burke LB. Clinical outcome assessments for clinical trials in children. In Pediatric Drug Development: Concepts and Applications (Eds. AE Mulberg, D Murphy, J Dunne and LL Mathis. John Wiley & Sons, Ltd, Hoboken, NJ, pp. 539-548.
- [Background] McLeod LD, Coon CD, Martin SA, Fehnel SE, Hays RD. Interpreting patient-reported outcome results: US FDA guidance and emerging methods. Expert Rev Pharmacoecon Outcomes Res. 2011 Apr;11(2):163-9. doi: 10.1586/erp.11.12. PMID 21476818
- [Background] Shroads AL, Langaee T, Coats BS, Kurtz TL, Bullock JR, Weithorn D, Gong Y, Wagner DA, Ostrov DA, Johnson JA, Stacpoole PW. Human polymorphisms in the glutathione transferase zeta 1/maleylacetoacetate isomerase gene influence the toxicokinetics of dichloroacetate. J Clin Pharmacol. 2012 Jun;52(6):837-49. doi: 10.1177/0091270011405664. Epub 2011 Jun 3. PMID 21642471
- [Background] Dunbar EM, Coats BS, Shroads AL, Langaee T, Lew A, Forder JR, Shuster JJ, Wagner DA, Stacpoole PW. Phase 1 trial of dichloroacetate (DCA) in adults with recurrent malignant brain tumors. Invest New Drugs. 2014 Jun;32(3):452-64. doi: 10.1007/s10637-013-0047-4. Epub 2013 Dec 3. PMID 24297161
- [Background] Shroads AL, Coats BS, McDonough CW, Langaee T, Stacpoole PW. Haplotype variations in glutathione transferase zeta 1 influence the kinetics and dynamics of chronic dichloroacetate in children. J Clin Pharmacol. 2015 Jan;55(1):50-5. doi: 10.1002/jcph.371. Epub 2014 Aug 6. PMID 25079374
- [Background] Stacpoole PW, Wright EC, Baumgartner TG, Bersin RM, Buchalter S, Curry SH, Duncan CA, Harman EM, Henderson GN, Jenkinson S, et al. A controlled clinical trial of dichloroacetate for treatment of lactic acidosis in adults. The Dichloroacetate-Lactic Acidosis Study Group. N Engl J Med. 1992 Nov 26;327(22):1564-9. doi: 10.1056/NEJM199211263272204. PMID 1435883
- [Background] Duncan GE, Perkins LA, Theriaque DW, Neiberger RE, Stacpoole PW. Dichloroacetate therapy attenuates the blood lactate response to submaximal exercise in patients with defects in mitochondrial energy metabolism. J Clin Endocrinol Metab. 2004 Apr;89(4):1733-8. doi: 10.1210/jc.2003-031684. PMID 15070938
- [Background] Stacpoole PW, deGrauw TJ, Feigenbaum AS, Hoppel C, Kerr DS, McCandless SE, Miles MV, Robinson BH, Tang PH. Design and implementation of the first randomized controlled trial of coenzyme CoQ(1)(0) in children with primary mitochondrial diseases. Mitochondrion. 2012 Nov;12(6):623-9. doi: 10.1016/j.mito.2012.09.005. Epub 2012 Sep 25. PMID 23022402
- [Background] Felitsyn NM, Henderson GN, James MO, Stacpoole PW. Liquid chromatography-tandem mass spectrometry method for the simultaneous determination of delta-ALA, tyrosine and creatinine in biological fluids. Clin Chim Acta. 2004 Dec;350(1-2):219-30. doi: 10.1016/j.cccn.2004.08.009. PMID 15530481
- [Background] Weber TA, Antognetti MR, Stacpoole PW. Caveats when considering ketogenic diets for the treatment of pyruvate dehydrogenase complex deficiency. J Pediatr. 2001 Mar;138(3):390-5. doi: 10.1067/mpd.2001.111817. PMID 11241048
- [Background] Shroads AL, Henderson GN, Cheung J, James MO, Stacpoole PW. Unified gas chromatographic-mass spectrometric method for quantitating tyrosine metabolites in urine and plasma. J Chromatogr B Analyt Technol Biomed Life Sci. 2004 Sep 5;808(2):153-61. doi: 10.1016/j.jchromb.2004.05.005. PMID 15261808
- [Background] Yan Z, Henderson GN, James MO, Stacpoole PW. Determination of dichloroacetate and its metabolites in human plasma by gas chromatography-mass spectrometry. J Chromatogr B Biomed Sci Appl. 1997 Dec 5;703(1-2):75-84. doi: 10.1016/s0378-4347(97)00404-0. PMID 9448064
- [Background] Martinelli D, Catteruccia M, Piemonte F, Pastore A, Tozzi G, Dionisi-Vici C, Pontrelli G, Corsetti T, Livadiotti S, Kheifets V, Hinman A, Shrader WD, Thoolen M, Klein MB, Bertini E, Miller G. EPI-743 reverses the progression of the pediatric mitochondrial disease--genetically defined Leigh Syndrome. Mol Genet Metab. 2012 Nov;107(3):383-8. doi: 10.1016/j.ymgme.2012.09.007. Epub 2012 Sep 10. PMID 23010433
- [Background] Shroads AL, Guo X, Dixit V, Liu HP, James MO, Stacpoole PW. Age-dependent kinetics and metabolism of dichloroacetate: possible relevance to toxicity. J Pharmacol Exp Ther. 2008 Mar;324(3):1163-71. doi: 10.1124/jpet.107.134593. Epub 2007 Dec 20. PMID 18096758
- [Background] Sperl W, Fleuren L, Freisinger P, Haack TB, Ribes A, Feichtinger RG, Rodenburg RJ, Zimmermann FA, Koch J, Rivera I, Prokisch H, Smeitink JA, Mayr JA. The spectrum of pyruvate oxidation defects in the diagnosis of mitochondrial disorders. J Inherit Metab Dis. 2015 May;38(3):391-403. doi: 10.1007/s10545-014-9787-3. Epub 2014 Dec 20. PMID 25526709
- [Background] Lehman, EL. Nonparametrics: Statistical methods Based on Ranks. (Page 173). Holden-Day, San Francisco, 1975.